CLINICAL TRIAL: NCT00918736
Title: Hyaluronans in the Treatment of Ankle Osteoarthritis
Brief Title: Efficacy of 3 Weekly Injections of Hyaluronate in Patients With Ankle Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Shu-Fen Sun, Kaohsiung Veteran General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NSC96-2314-B-075B-006
Record Dates: First submitted 2009-03-16; First posted 2009-06-11 (Estimated); Results first posted 2009-06-11 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Osteoarthritis
Keywords: Ankle joint; Balance; Hyaluronic acid; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hyaluronate injection (Experimental): All patients with unilateral ankle OA received 3 weekly intraarticular injections of 2 ml sodium hyaluronate (Hyalgan) into the ankle joints.
  Interventions: Drug: sodium hyaluronate

INTERVENTIONS:
Drug: sodium hyaluronate — 3 weekly intraarticular injections of 2 ml sodium hyaluronate (Hyalgan) into the ankle joints.

SUMMARY:
The aim of this study was to investigate the efficacy and safety of three weekly intraarticular injections of Hyaluronate (HA) in patients with unilateral ankle Osteoarthritis (OA).

DETAILED DESCRIPTION:
Viscosupplementation with 3 to 5 weekly hyaluronate injections is a well-established treatment option in knee osteoarthritis. Previous studies reported that five weekly hyaluronate injections were safe and effective for the treatment of ankle osteoarthritis. However, the effect of three weekly injections has rarely been investigated. Besides, no study to date has assessed whether balance function would change after HA injections in patients with ankle OA. The purpose of this study was to evaluate the efficacy and safety of three weekly injections of sodium hyaluronate (Hyalgan) in patients with unilateral ankle osteoarthritis. Pain, physical function and balance will be assessed as parameters for the effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* were 18 years of age or older, reported unilateral ankle pain for at least 6 months and had either reported no significant benefit from conservative treatment (rest, physical therapy, orthoses or pain medications etc.) or were unable to tolerate side effects of medications
* ankle radiographs taken within 6 months were equivalent to grade 2 or 3 according to the Kellgren-Lawrence grading system (grade 2, definite osteophytes and possible narrowing of joint space; grade 3, moderate multiple osteophytes, definite narrowing of joint space, some sclerosis and possible deformity of bone contour)22
* had a current total AOS score (described below) of > 3 and < 9 (possible range, 0-10)
* were normally active, not bedridden or confined to a wheelchair, and were able to walk 30 meters without the aid of a walker, crutches or cane
* were willing to discontinue all nonsteroidal anti-inflammatory drugs (NSAIDs) or other analgesic medication (except for rescue medication) for the duration of the study
* did not receive physical therapy or trial of shoe modifications or orthotics during the study period

Exclusion Criteria:

* pregnant and lactating women
* bilateral ankle OA requiring treatment of both ankles
* chronic ankle instability
* lower leg trauma other than within the ankle
* previous orthopedic surgery on the spine, hip or knee
* presence of active joint infections of foot or ankle
* previous surgery or arthroscopy on the ankle within 12 months
* intraarticular steroid or HA injection in the treated ankle within the past 6 months
* treatment with anticoagulants or immunosuppressives
* history of rheumatoid arthritis, gout, or any other inflammatory arthropathy
* history of avian protein allergy
* presence of other comorbidity (neoplasm, diabetes mellitus, paresis, recent trauma, etc) or poor health status that would interfere with the clinical assessments during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Fen Sun, MD, Principal Investigator — Veterans General Hospital, Kaohsiung, Taiwan
Locations (1):
- Department of Physical Medicine and Rehabilitation, Veterans General Hospital, Kaohsiung, Taiwan, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Salk RS, Chang TJ, D'Costa WF, Soomekh DJ, Grogan KA. Sodium hyaluronate in the treatment of osteoarthritis of the ankle: a controlled, randomized, double-blind pilot study. J Bone Joint Surg Am. 2006 Feb;88(2):295-302. doi: 10.2106/JBJS.E.00193. PMID 16452740
- [Background] Sun SF, Chou YJ, Hsu CW, Hwang CW, Hsu PT, Wang JL, Hsu YW, Chou MC. Efficacy of intra-articular hyaluronic acid in patients with osteoarthritis of the ankle: a prospective study. Osteoarthritis Cartilage. 2006 Sep;14(9):867-74. doi: 10.1016/j.joca.2006.03.003. Epub 2006 Apr 24. PMID 16635582
- [Background] Cohen MM, Altman RD, Hollstrom R, Hollstrom C, Sun C, Gipson B. Safety and efficacy of intra-articular sodium hyaluronate (Hyalgan) in a randomized, double-blind study for osteoarthritis of the ankle. Foot Ankle Int. 2008 Jul;29(7):657-63. doi: 10.3113/FAI.2008.0657. PMID 18785414

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty patients fulfilled the inclusion criteria and consented to take part in this study.
Pre-assignment Details: One patient withdrew his consent and one had a fear of injection prior to receiving the first injection. Two patients withdrew from the study before the third injection (one because of an unrelated intercurrent illness and one moving to another city).
Period: Overall Study
Arm/Group | Hyaluronate Injection
Started | 50 (October, 2007)
Completed | 46 (October, 2008)
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Hyaluronate Injection
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 51.7 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 22
Region of Enrollment [Number; unit: participants]
  Taiwan | 50

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Ankle Osteoarthritis Scale (AOS) Score at 6 Months
Description: The AOS is a patient-rated, validated outcome measure that includes nine items on a pain subscale and nine items on a disability subscale. Using the AOS, a score of 0 represent no pain or disability and 10 represent worst pain or disability imaginable
Time Frame: baseline and 6 months
Population: The statistical analysis was done on completers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyaluronate Injection
Number analyzed (Participants) | 46
score on a scale | 2.3 (1.7)
Statistical Analysis 1: Comparison: Hyaluronate Injection; Previous report using 5 weekly injections, mean AOS score reduction is 2.6 with the SD of 1.8 in 75 patients. To test whether AOS reduction would be > 1 using pair t-test after 3 weekly injections, investigators need > 42 patients to give > 90% power to reject the null hypothesis-mean AOS score reduction <1 at 6 months, given that both the mean and standard deviation of AOS score reduction equal to 2. Considering possible dropout of participants, investigators decide to include 50 patients; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: The American Orthopedic Foot and Ankle Society (AOFAS) Ankle/Hindfoot Score
Description: The American Orthopedic Foot and Ankle Society (AOFAS) ankle/hindfoot score is a 100-point scale that devotes 40 points to pain, 50 points to function and 10 points to alignment. The maximum score of 100 points denotes no pain and normal function and alignment
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2009-10
Measure: Mean (Standard Deviation); unit: point

3. Secondary Outcome: Ankle Sagittal Range of Motion
Description: Ankle sagittal ROM is the sum of ankle dorsiflexion and plantar flexion angles.
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2009-09
Measure: Mean (Standard Deviation); unit: degree

4. Secondary Outcome: Four Clinical Balance Tests
Description: Single-leg stance test (SLS),The Functional Reach Test (FRT),Timed " Up-and-Go" test (TUG) ,Berg Balance Scale (BBS)
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2009-09
Measure: Mean (Standard Deviation); unit: sec

5. Secondary Outcome: the Level of Global Satisfaction Based on a 7-point Categorical Scale
Description: The rating was based on a 7-point categorical scale weighted from completely satisfied, satisfied, somewhat satisfied, no change, somewhat unsatisfied, unsatisfied to completely unsatisfied.
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2009-10
Measure: Number; unit: participants

6. Secondary Outcome: Systemic and Local Adverse Events Recording
Description: he occurrence of systemic and local adverse events, defined as any unwanted events whether it was thought to be related to the study drugs or not, were recorded on a diary card
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2009-10
Measure: Number; unit: participants

7. Secondary Outcome: Rescue Acetaminophen Consumption
Description: The use of all analgesic medication during the study period was recorded on a diary card by the patient.
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2009-10
Measure: Mean (Standard Deviation); unit: tablets

ADVERSE EVENTS:
Arm/Group | Hyaluronate Injection
Serious Adverse Events (participants affected / at risk) | 0
Other Adverse Events (participants affected / at risk) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 8.7% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Hyaluronate Injection
brief post injection pain (Skin and subcutaneous tissue disorders) | 3/3 (3)
local pruritis (Skin and subcutaneous tissue disorders) | 1/1 (1)

LIMITATIONS AND CAVEATS:
One limitation includes the absence of a control group, thus the placebo effects associated with joint injections were not investigated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes